CLINICAL TRIAL: NCT05577741
Title: Effect of the Enriched Environment on the Risk of Relapse: Clinical Study Combining Physical Activity With Mindfulness in Virtual Reality
Brief Title: Effect of the Enriched Environment on the Risk of Relapse
Acronym: ENVELMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01156-37
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alcoholic Relapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Patients complete a measurement session at inclusion visit (Day 1). These measures include an assessment of explicit and implicit craving, a measure of mindfulness skills and a measure of the perceived richness (in stimuli) of daily environment. After inclusion visit, patients randomized in the interventional group will have 6 sessions of enriched environment (from Day 2 to Day 9).
  The enriched environment includes:
  * the multisensory virtual reality pod offers sessions of 20 minutes of mindfulness in immersive situations. Some immersive situations are relaxing and others trigger cues in order to improve craving management;
  * the cognitive bike offers training sessions of 20 minutes. The patient pedals while using a touch pad with cognitive training games. This simultaneously stimulate motor skills and cognition by means of bicycle-game coupling.
  A second measurement session takes place at Day 10. Alcoholic relapse is then evaluated at two weeks, one month and 3 months.
  Interventions: Behavioral: Multisensory virtual reality pod (SENSIKS©); Behavioral: Cognitive bike (Vélo-cognitif®); Other: Standard treatment
- Control Group (Active Comparator): Patients complete a similar measurement session to the intervention arm, that include psychological tasks and questionnaires at inclusion visit (Day 1). After inclusion visit, patients randomized in the control group wil received the standard of care.
  A second measurement session takes place at Day 10. Alcoholic relapse is then evaluated at two weeks, one month and 3 months.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Multisensory virtual reality pod (SENSIKS©) — Six sessions of 20 minutes of mindfulness.
  Arms: Interventional Group
Behavioral: Cognitive bike (Vélo-cognitif®) — Six sessions of 20 minutes of cognitive bike (pedal + cognitive games).
  Arms: Interventional Group
Other: Standard treatment — Standard of care treatment

SUMMARY:
This clinical study investigates the effects of enriched environment on the risk of relapse in alcoholic patients.

135 patients hospitalized for an alcoholic addiction will be recruited and randomized in two groups: one group will receive standard of care, the other group will receive a treatment with enriched environment.

The enriched environment consists of six sessions of virtual reality (20 minutes) in a multi-sensory pod and six sessions (20 minutes) of bike activity with cognitive tasks while pedalling.

The multi-sensory virtual reality pod allows mindfulness practice and allows patients to be in immersive situations that may trigger cues in order to help them in craving management.

The bike consists in the combination of a pedal set and a touch pad on which cognitive training games are offered. This tool thus makes it possible to simultaneously stimulate motor skills and cognition by means of bicycle-game coupling.

Patients are then followed during 3 months and a half.

ELIGIBILITY:
Inclusion Criteria:

* Any patient hospitalized at the Henri Laborit Hospital for alcohol addiction, on an opened unit for at least 48 hours;
* Woman or man aged between 18 and 65 inclusive
* Severe alcohol use disorder according to the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders
* Benefit from social security or benefit from it through a third party in accordance with French law on research involving the human person
* Have signed the informed consent form after receiving written information.

Exclusion Criteria:

* Disabling cognitive disorders
* Cardiological pathologies that could compromise the participation of patients, detected by an ECG.
* Advanced pulmonary, renal, and hepatic diseases, or any unstable and serious medical conditions that could compromise the patient's participation in the study, subject to the judgment of the doctor
* Hypertension
* Ataxia
* Uncompensated and unstable psychiatric pathology
* Susceptibility to cybersickness
* Pregnant or breastfeeding woman
* Simultaneous participation in another trial
* Any other current addiction, except addiction to tobacco and benzodiazepines
* Employee of the investigator or of the clinical study site
* Patients protected by law
* People not covered by state health insurance
* Patients who in the opinion of the investigator are unable to complete the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Alcoholic relapse | 2 weeks
  Relapse at 2 weeks (after Day 10), defined by the consumption of at least 5 glasses per occasion, or by consumption at least 5 times a week, assessed by the Time Line Follow Back, a beathalyser or a significant increase in Carbohydrate Deficient Transferrin and Gamma-GT.
  We will consider a relapse to have occurred if at least one of the three indicators points to a relapse: 1) if in the TLFB the patient indicates consumption of at least 5 times per week or at least 5 drinks per occasion; 2) if there is a significant increase in CDT and GGT since the D10 blood test, and 3) If the breathalyser is positive. We will consider patients as non-relapsers if none of these indicators (TLFB, CDT and GGT, breathalyzer) is positive.

SECONDARY OUTCOMES:
Alcoholic relapse | 1 month
  Relapse at 1 month (after Day 10), defined by the consumption of at least 5 glasses per occasion, or by consumption at least 5 times a week
Alcoholic relapse | 3 months
  Relapse at 3 months (after Day 10), defined by the consumption of at least 5 glasses per occasion, or by consumption at least 5 times a week
Explicit craving | Day 10
  The effect of intervention on explicit craving, assessed by the Obsessive Compulsive Drinking Scale and the cue craving induction protocol.
Implicit craving | Day 10
  The effect of intervention on implicit craving, assessed by an Implicit Association Test, a test of the seeking for alcohol-related stimuli, and a visual research test for alcohol-related stimuli (eye-tracking)
Mindfulness skills | Day 10
  The effect of intervention on mindfulness skills, assessed by a questionnaire (Five Facets Mindfulness Questionnaire -15)
Perception of the richness of the daily environment | Day 10
  The effect of the intervention on the perceived richness of the daily environment, assessed by a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available (including data dictionaries) to researchers upon reasonable request, beginning 9 months following article publication (no end date). All the deidentified individual participant data collected during the trial, study protocol, statistical analysis plan, informed consent form, and analytic code will be shared. Data will be available for any purpose by writing a request to lila.barillot@uiv-poitiers.fr.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months following article publication (no end date)
Access Criteria: Researchers upon reasonable request

REFERENCES:
- [Derived] Barillot L, Chauvet C, Besnier M, Jaafari N, Solinas M, Chatard A. Effect of environmental enrichment on relapse rates in patients with severe alcohol use disorder: protocol for a randomised controlled trial. BMJ Open. 2023 May 12;13(5):e069249. doi: 10.1136/bmjopen-2022-069249. PMID 37173113